CLINICAL TRIAL: NCT04428372
Title: MAnnitol for Blood Pressure Stability in HemoDialysis (MAP-HD)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Finnian McCausland, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019P003681
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Hemodialysis Complication; Hemodynamic Instability
Keywords: hemodialysis
MeSH Terms: interventions — Mannitol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mannitol (Experimental): intravenous 20% mannitol, 0.25g/kg/hour (maximum 25g/hour; maximum 75g per session; maximum volume 375mL/session) as a continuous infusion during dialysis
  Interventions: Drug: Mannitol
- Placebo (Placebo Comparator): 0.9% saline at a rate of 1.25mL/kg/hour (maximum volume 375mL) as a continuous infusion during dialysis
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Mannitol — Hypertonic mannitol infusion
  Arms: Mannitol
Drug: 0.9% saline — Normal saline 'placebo' arm
  Arms: Placebo

SUMMARY:
This proposal will measure the effects of mannitol administration versus placebo in hypotensive-prone, adult, maintenance hemodialysis patients with respect to changes in patient symptoms and blood pressure stability.

DETAILED DESCRIPTION:
A randomized crossover trial of hypertonic mannitol vs. placebo in IDH-prone participants will be performed over a 4-week period to determine the effect on:

* Patient symptoms
* The magnitude of intra-dialytic hypotension

The hypothesis to be tested is that the use of hypertonic mannitol will result in fewer adverse symptoms and less decline in intra-dialytic BP, compared with the use of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Maintenance HD (>90 days)
* Age ≥18y
* Thrice-weekly HD
* IDH-prone (defined as nadir intra-dialytic SBP <100 mmHg in ≥30% of sessions in the prior 4 weeks)
* Hematocrit>21%
* Written informed consent

Exclusion Criteria:

* Acute myocardial infarction or stroke within one month
* Pre-HD serum potassium >6.5 mmol/L in last 4 weeks
* Pregnancy
* Institutionalized individuals
* Life expectancy <2 months
* Planned renal transplant within 2 months
* Active enrollment in another interventional trial
* Known allergy to mannitol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Patient Symptoms | 4 weeks
  Comparison of average patient symptom score during mannitol arm using dialysis symptom index compared with the average score during the placebo arm (scale 0-150; higher scores worse)

SECONDARY OUTCOMES:
Patient Symptoms | 4 weeks
  Comparison of average patient symptom score during mannitol arm using modified Edmonton symptom assessment system compared with the average score during the placebo arm (scale 0-100; higher scores worse)
Patient Symptoms | 4 weeks
  Comparison of average patient symptom score during mannitol arm using SMAART HD questionnaire compared with the average score during the placebo arm (scale 0-60 on 12-questions, higher scores worse)
Intra-dialytic hypotension | 4 weeks
  Comparison of change in average intra-dialytic systolic blood pressure change during mannitol arm, compared with during the placebo arm

CONTACTS AND LOCATIONS:
Overall Officials: Finnian R Mc Causland, MBBCH, MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Modest sized single-center study with no plan to share individual participant data